CLINICAL TRIAL: NCT04509843
Title: Impact of Socioeconomic Status and Oral Hygiene Practice on Periodontal Health of Egyptian Adults: A Hospital Based Cross-sectional Study
Brief Title: Impact of Socioeconomic Status and Oral Hygiene Practice on Periodontal Health of Egyptian Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Alsayed Mohamed Alsayed Alsadany (Other)
Responsible Party: Sponsor-Investigator, Alsayed Mohamed Alsayed Alsadany, Principal Investigator, Cairo University
Organization: Cairo University (Other)
Other Study IDs: 3-4-20
Record Dates: First submitted 2020-07-20; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-07

CONDITIONS: Periodontal Health
MeSH Terms: interventions — Social Class

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: socioeconomic status — it is a cross-sectional study for assessment the impact of socioeconomic status on periodontal health through using a definite scale mentioned in the protocol related to the middle east people.

SUMMARY:
evaluation the relationship between the socioeconomic status and periodontal health of Egyptian adults.

DETAILED DESCRIPTION:
It is a cross-sectional study for evaluation and assessment of periodontal health, socioeconomic status and oral hygiene measurements among Egyptian adults recruiting from the outpatient clinic and the payed treatment clinics at faculty of Dentistry, Cairo University.

The faculty of Dentistry, Cairo University is an open public facility, a tertiary healthcare and a referral center.

ELIGIBILITY:
Inclusion Criteria:

* -Patients whose age is 18-70 years old recruiting from the outpatient clinic and the payed clinic
* Provide informed consent.

Exclusion Criteria:

* Patients having problem in opening their mouth or undergoing intermaxillary fixation where oral examination will not be possible.
* Patients diagnosed with psychiatric problems or intoxicated with alcohol or drugs.
* pregnant patients.
* patients undergoing orthodontic treatment.
* patients who had undergone periodontal treatment over the past six months.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients will be recruited in a consecutive manner from the outpatient Diagnostic center, Faculty of Dentistry, Cairo University.
Sampling Method: Probability Sample
Enrollment: 456 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Periodontal health | "through study completion, an average of 1 year"
  Recently, definition of periodontal health has been developed dramatically from just the absence of a disease to a state around a stable periodontium (Lang and Bartold, 2018) that functions in comfort in an individual with psychological and social well-being about their mouth (Mariotti and Hefti, 2015). Based on this, biological, environmental, systemic, social, economic and psychological factors can affect periodontal health in different ways.
  Periodontal examination using the community periodontal index (CPI) will be done for all of the participants to assess the status of periodontal condition. The CPITN criteria used in this study will be as follows: score 0 = healthy periodontium with no sign of periodontal disease, score 1= gingival bleeding on probing, 2=calculus deposits, 3=pockets 4-5mm (shallow pockets), 4=pockets 6mm or deeper (deep pockets) and X =excluded sextants.
periodontal disease | through study completion, an average of 1 year
  Periodontal diseases have been categorized in a new framework: stage I to VI of periodontitis based on severity, complexity of management with additional described extent as localized or generalized. Grade A to C of periodontitis related to the progression rate of the disease as slow, moderate and rapid with grade modifiers. The seriousness and the complexity of the disease are greater as the grade increases within each stage.(Tonetti, Greenwell and Kornman, 2018).
  Information on loss of attachment (CAL) will be collected from the same index teeth using CPI modified system. The two molars in each posterior sextant are paired for recording and if one is missing there is no replacement. If no index tooth is present in a sextant qualifying for examination, all teeth present in that sextant are examined and the highest score is recorded as the score for the sextant WHO.

SECONDARY OUTCOMES:
Impact of sociodemographic factors on periodontal health | through study completion, an average of 1 year
  Patient-centered approaches turned to be more popular, which increased the attention to the effects of different human health situations on periodontal health through the concept that the way in which an individual' lives may produce behavioural patterns that are either beneficial or determinable to health including socioeconomic status.
  Social class will be classified according to following socioeconomic status scale for health research in Egypt into low, moderate and high socioeconomic subgroups described by El-Gilany et al. (El-Gilany, El-Wehady and El-Wasify, 2012) This scale includes 7 domains with a total score of 84. Socioeconomic level: to be classified into very low, low, middle and high levels depending on the quartiles of the score calculated.
impact of periodontal practice on periodontal health | through study completion, an average of 1 year
  (Lertpimonchai et al., 2017) concluded that fair to poor oral hygiene measures especially irregular tooth brushing increases the risk of periodontal disease by two to five folds in conjunction with low frequency tooth brushing which was conducted in a systematic-review with severe forms of periodontal diseases.
  periodontal practice will be addressed via several questions that evaluate the self-care practices of tooth brushing, flossing, mouth rinsing in recent one year, scaling in recent five years, and how to alleviate gingival bleeding if there is.The questionnaire will be filled through a face-to-face personal interview with the patient using simple, short, easily comprehended questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
i will share final statistical results.